CLINICAL TRIAL: NCT04570488
Title: Predicting Favorable Outcomes in Hospitalized Covid-19 Patients
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: PAU COVID19
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: COVID; Corona Virus Infection; Adverse Event
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Quality improvement - Display: Display of risk score/ colored flag in Epic patient list column; will be viewable to all frontline workers
  Interventions: Other: EPIC risk score display
- No Display: No display ("hidden") of risk score/ colored flag in Epic patient list column; not viewable to all frontline workers

INTERVENTIONS:
Other: EPIC risk score display — Display of risk score/ colored flag in Epic patient list column
  Groups: Quality improvement - Display

SUMMARY:
Testing use of predictive analytics to predict which COVID-19+ patients are at low risk for an adverse event (ICU transfer, intubation, mortality, hospice discharge, re-presentation to the ED, oxygen requirements exceeding nasal cannula at 6L/Min) in the next 96 hours

DETAILED DESCRIPTION:
To assess if display of low risk of adverse event in EPIC can safely reduce length of stay and plan for discharge.

ELIGIBILITY:
Inclusion Criteria: Adult hospitalized COVID19+ patients predicted to have no adverse event at 96 events with a threshold at 90% PPV, with at least one low risk during their admission who are discharged alive and have not been in the ICU

Exclusion Criteria: Age < 18 years not hospitalized for COVID19+.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hospitalized COVID19+ patients predicted to have no adverse event at 96 events with a threshold at 90% PPV, with at least one low risk during their admission who are discharged alive and have not been in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 1415 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Reduction in days from first low-risk score to discharge | 96 Hours
  Reduction in days from first low-risk score to discharge

SECONDARY OUTCOMES:
Reduction in length of stay (LOS) | 96 hours
  Reduction in LOS for green patients that have not been in the ICU
Reduction in GTD vs. LOS | 96 hours
  Reduction in GTD vs. LOS for all green patients discharged alive vs all patients discharged alive
No change in 30 day re-ED presentation or hospital admission rate for cohort | 96 hours
  No change in 30 day re-ED presentation or hospital admission rate for cohort

OTHER OUTCOMES:
Re-presentation to ED | 96 hours
Readmission to hospital | 96 hours
Mortality | 96 hours
Postdischarge mortality | 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Austrian, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Major VJ, Jones SA, Razavian N, Bagheri A, Mendoza F, Stadelman J, Horwitz LI, Austrian J, Aphinyanaphongs Y. Evaluating the Effect of a COVID-19 Predictive Model to Facilitate Discharge: A Randomized Controlled Trial. Appl Clin Inform. 2022 May;13(3):632-640. doi: 10.1055/s-0042-1750416. Epub 2022 Jul 27. PMID 35896506